CLINICAL TRIAL: NCT00363090
Title: Alemtuzumab and CHOP Chemotherapy for Aggressive Histology Peripheral T Cell Lymphomas: A Multi-Centre Phase I and II Study
Brief Title: Alemtuzumab and Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage II, Stage III, or Stage IV T-Cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Sunnybrook Regional Cancer Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000491451; TSRCC-164-2006
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Alemtuzumab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Flow Cytometry

INTERVENTIONS:
Biological: alemtuzumab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Other: flow cytometry
Other: pharmacological study

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from growing. Giving alemtuzumab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of alemtuzumab when given together with combination chemotherapy and to see how well they work in treating patients with newly diagnosed aggressive stage II, stage III, or stage IV T-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the safety and dose-limiting toxicities of alemtuzumab in combination with cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (CHOP) chemotherapy in patients with newly diagnosed, stage II-IV aggressive peripheral T-cell non-Hodgkin's lymphoma.
* Measure the pharmacokinetics of alemtuzumab using different subcutaneous doses and schedules to determine the dose with the highest achievable drug levels with acceptable toxicities worthy of further investigation.

Secondary

* Determine the efficacy of alemtuzumab in combination with CHOP chemotherapy using escalating doses and 2 different drug schedules, as defined by overall response rate, progression-free survival, and overall survival.
* Measure the effects of this regimen on T-cell reconstitution and cytomegalovirus reactivation.

OUTLINE: This is a multicenter, phase I, dose-escalation study of alemtuzumab followed by an open-label, phase II study.

* Phase I: Patients receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Patients also receive alemtuzumab subcutaneously (SC) on day 1 OR on days 1, 8, and 15. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of alemtuzumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive CHOP chemotherapy and alemtuzumab (at the MTD determined in phase I) as in phase I (on the most effective regimen).

Patients undergo blood collection at baseline, periodically during study treatment, and after completion of study treatment for pharmacokinetics and other correlative studies. Samples are examined for presence of cytomegalovirus antigen and by flow cytometry for B- and T-cell quantification.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 84 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive peripheral T-cell non-Hodgkin's lymphoma (NHL), including the following nodal or extranodal subtypes:

  * Nodal:

    * Angioimmunoblastic lymphadenopathy
    * ALK 1-negative anaplastic large cell NHL
    * Peripheral T-cell lymphoma not otherwise specified
  * Extranodal:

    * Hepatosplenic NHL
    * Enteropathy-associated NHL
    * Panniculitic NHL
* Stage II-IV disease
* Newly diagnosed, CD52+ disease
* Measurable or evaluable disease
* No known CNS involvement with lymphoma
* No nasal natural killer T-cell NHL

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 4 months
* Absolute neutrophil count ≥ 1,000/mm³*
* Platelet count ≥ 75,000/mm³*
* Hemoglobin ≥ 8.5 g/dL*
* Bilirubin < 2.0 mg/dL
* Alkaline phosphatase ≤ 2 times upper limit of normal (ULN)
* AST or ALT < 2 times ULN
* Creatinine < 1.5 mg/dL*
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to any of the study drugs
* No serious illnesses that would preclude compliance with study requirements
* No known HIV positivity
* No other preexisting immunodeficiency (e.g., post-organ transplant)
* No other malignancy within the past 5 years except cervical carcinoma in situ or nonmelanoma skin cancer NOTE: *Unless directly attributable to NHL

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

  * Up to 7 days of prednisone preceding initiation of chemotherapy allowed
* No other concurrent chemotherapy, radiotherapy, or immunotherapy
* No other concurrent corticosteroids except dexamethasone used as an antiemetic for a brief period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity as assessed by NCI Common Toxicity Criteria Version 3.0
Safety
Dose-limiting toxicities
Pharmacokinetics of alemtuzumab

SECONDARY OUTCOMES:
Efficacy as assessed by clinical, radiologic, pathologic, and laboratory measurements
Overall response rate
Progression-free survival
Overall survival
Effects of treatment on T- and B-cell reconstitution by flow cytometry at baseline and at 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (5):
- Canada (5):
  - St. Paul's Hospital at Providence Health Care - Vancouver, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario